CLINICAL TRIAL: NCT02610010
Title: Intensity-modulated Radiotherapy With or Without Concurrent Chemotherapy for Stage II Nasopharyngeal Carcinoma: a Phase 3 Non-inferior Multicenter Randomized Controlled Trial
Brief Title: Intensity-modulated Radiotherapy With or Without Concurrent Chemotherapy for Stage II Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-FXY-066-Dept. of RT
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: NPC; concurrent chemotherapy; IMRT; stage II
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMRT alone (Experimental): Intensity-modulated radiotherapy without cisplatin-based concurrent chemotherapy
  Interventions: Radiation: Intensity-modulated radiotherapy
- IMRT plus concurrent chemotherapy (Active Comparator): Intensity-modulated radiotherapy with cisplatin-based concurrent chemotherapy
  Interventions: Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 100 mg/m² every 3 weeks for 3 cycles during radiotherapy.
  Other Names: DDP
  Arms: IMRT plus concurrent chemotherapy
Radiation: Intensity-modulated radiotherapy — Intensity-modulated radiotherapy

SUMMARY:
A prior phase III randomized trial showed considerable survival benefit from the combined treatment of cisplatin-based concurrent chemotherapy and two-dimensional conventional radiotherapy (2DCRT) for patients with stage II (the Chinese 1992 staging system) nasopharyngeal carcinoma. However, since intensity-modulated radiotherapy (IMRT) was known to be superior to 2DCRT in local control, progression free survival and even overall survival, it is a pivotal question whether stage II [T1N1M0 and T2N0-1M0, based on the 2010 International Union against Cancer/American Joint Committee on Cancer (UICC/AJCC) staging system] patients can still obtain significant benefit from the additional concurrent chemotherapy in the IMRT era.

The investigators' retrospective study (PMID:26528755 ) indicated that low risk nasopharyngeal carcinoma (T1N1M0, T2N0-1M0 or T3N0M0, the 2010 UICC/AJCC staging system) patients who underwent IMRT could not benefit from cisplatin-based concurrent chemotherapy. Therefore, the investigators perform this randomized controlled trial to address this question, on a prudent assumption that IMRT alone was not inferior to IMRT plus concurrent chemotherapy in stage II patients.

DETAILED DESCRIPTION:
Eligible patients are randomly assigned to receive intensity-modulated radiotherapy (IMRT) alone or IMRT plus concurrent chemotherapy. IMRT is given as 2.0-2.30 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor. Concurrent chemotherapy consisted of cisplatin 100 mg/m² every 3 weeks for 3 cycles. The primary endpoint is overall survival (OS). Secondary end points include failure-free survival(FFS), locoregional relapse-free survival (LRFS), distant metastasis-free survival (DMFS), toxic effects and quality of life. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologically confirmed non-keratinizing (WHO 1991) nasopharyngeal carcinoma.
* Tumor staged as T1N1M0 or T2N0-1M0 (the 2010 UICC/AJCC staging system).
* Karnofsky scale (KPS) ≥ 70.
* Adequate marrow: leucocyte count ≥ 4×10E9/L, hemoglobin ≥ 110g/L and platelet count ≥ 100×10E9/L.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and bilirubin ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN.
* Adequate renal function: creatinine clearance ≥ 60 ml/min or creatinine ≤ 1.5×ULN.
* Patients must give written informed consent.

Exclusion Criteria:

* Prior malignancy, except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended radiotherapy volume).
* Prior radiotherapy, chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Estimated)
Dates: Start 2015-11; Primary Completion 2022-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Two year

SECONDARY OUTCOMES:
failure-free survival | two year
distant metastasis-free survival | two year
locoregional relapse-free survival | two year
Number of participants with treatment-related acute adverse events as assessed by CTCAE v4.0 | two months
quality of life assessing by questionnaires | through study completion, an average of 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Yun Xie, M.D., Principal Investigator — Sun Yat-sen University Cancer Center,Guangzhou, Guangdong, China
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang LN, Gao YH, Lan XW, Tang J, Su Z, Ma J, Deng W, OuYang PY, Xie FY. Propensity score matching analysis of cisplatin-based concurrent chemotherapy in low risk nasopharyngeal carcinoma in the intensity-modulated radiotherapy era. Oncotarget. 2015 Dec 22;6(41):44019-29. doi: 10.18632/oncotarget.5806. PMID 26528755
- [Background] Su Z, Mao YP, Tang J, Lan XW, OuYang PY, Xie FY. Long-term outcomes of concurrent chemoradiotherapy versus radiotherapy alone in stage II nasopharyngeal carcinoma treated with IMRT: a retrospective study. Tumour Biol. 2016 Apr;37(4):4429-38. doi: 10.1007/s13277-015-4266-5. Epub 2015 Oct 25. PMID 26499947
- [Background] Chen QY, Wen YF, Guo L, Liu H, Huang PY, Mo HY, Li NW, Xiang YQ, Luo DH, Qiu F, Sun R, Deng MQ, Chen MY, Hua YJ, Guo X, Cao KJ, Hong MH, Qian CN, Mai HQ. Concurrent chemoradiotherapy vs radiotherapy alone in stage II nasopharyngeal carcinoma: phase III randomized trial. J Natl Cancer Inst. 2011 Dec 7;103(23):1761-70. doi: 10.1093/jnci/djr432. Epub 2011 Nov 4. PMID 22056739
- [Background] Lai SZ, Li WF, Chen L, Luo W, Chen YY, Liu LZ, Sun Y, Lin AH, Liu MZ, Ma J. How does intensity-modulated radiotherapy versus conventional two-dimensional radiotherapy influence the treatment results in nasopharyngeal carcinoma patients? Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):661-8. doi: 10.1016/j.ijrobp.2010.03.024. Epub 2010 Jul 17. PMID 20643517
- [Background] Zhang MX, Li J, Shen GP, Zou X, Xu JJ, Jiang R, You R, Hua YJ, Sun Y, Ma J, Hong MH, Chen MY. Intensity-modulated radiotherapy prolongs the survival of patients with nasopharyngeal carcinoma compared with conventional two-dimensional radiotherapy: A 10-year experience with a large cohort and long follow-up. Eur J Cancer. 2015 Nov;51(17):2587-95. doi: 10.1016/j.ejca.2015.08.006. Epub 2015 Aug 26. PMID 26318726
- [Background] Peng G, Wang T, Yang KY, Zhang S, Zhang T, Li Q, Han J, Wu G. A prospective, randomized study comparing outcomes and toxicities of intensity-modulated radiotherapy vs. conventional two-dimensional radiotherapy for the treatment of nasopharyngeal carcinoma. Radiother Oncol. 2012 Sep;104(3):286-93. doi: 10.1016/j.radonc.2012.08.013. Epub 2012 Sep 17. PMID 22995588